CLINICAL TRIAL: NCT02915640
Title: Remote Technology for Paediatric Patient Assessment, Stabilization and Triaging Prior to Paediatric Inter-facility Transportation: A Feasibility Study
Brief Title: Use of a Mobile Remote Device to Optimize Pediatric Inter-facility Transportation: A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Tanya Holt, Clinical Assistant Professor, University of Saskatchewan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PITROBOT-1
Record Dates: First submitted 2016-09-21; First posted 2016-09-27 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Acute Disease
MeSH Terms: conditions — Acute Disease | interventions — Remote Sensing Technology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remote technology (Experimental): Remote technology will be used for an initial patient assessment after being contacted by phone from the peripheral center to transfer an acutely ill pediatric patient as assessed by the referral centre care provider.
  Interventions: Other: Remote technology
- Control (No Intervention): A Nurse Practitioner or General Practitioner from a remote site has a pediatric acute care referral and arranges a transportation. There is an initial call to obtain a patient history, to provide advice to the remote caregiver to initiate specific therapies and to mobilize the specialized team to the patient.

INTERVENTIONS:
Other: Remote technology — Utilization of remote technology versus not using remote technology when triaging and managing pediatric patients in remote settings prior to pediatric specialized inter-facility transportation.
  Arms: Remote technology

SUMMARY:
This study compares the utilization of remote technology versus not using remote technology when triaging and managing pediatric patients in remote settings prior to pediatric specialized inter-facility transportation.

DETAILED DESCRIPTION:
Paediatric Specialized Inter-facility transport utilizes specialized teams usually made up of a respiratory therapist, paediatric critical care nurse, and paediatric intensivist as medical control. When a Nurse Practitioner or General Practitioner from a remote site has a paediatric acute care referral and wants to arrange transportation there is an initial call at which point there are two priorities: first is obtain a patient history and then provide advice to the remote caregiver to initiate specific therapies; second is to mobilize the specialized team to the patient. The period of time between giving initial advice while dispatching the team and the time when the team arrives, can often be a vulnerable period for the remote caregiver as well as the patient. The ability to directly visualize and assess the patient during this time, as well as assist the specialized team once they arrive may provide improvement in safety and care of the patient. It may also improve triaging and may make the stabilization and departure time more efficient.

Remote technology will be used for an initial patient assessment after being contacted by phone from the peripheral centre to transfer an acutely ill paediatric patient as assessed by the referral centre care provider. After assessment the patient will be triaged to either remain in the local community, transferred to a regional hospital that provides paediatric acute care (Prince Albert), or be transported to Royal University Hospital in Saskatoon for tertiary care. Data to be collected includes:

* Duration of time from the beginning of the initial phone call to the first therapeutic intervention
* Time to stabilization
* Time to decision for disposition
* The duration of contact with the health care provider and the patient
* Number of scheduled follow-up contacts for a specific patient within 24 hours
* Number of times the referring centre re-consults
* Of the patients who triaged to stay in the local community how many were transported to the tertiary care centre within 24hrs
* How many patients who arrived at the tertiary care centre were discharged within 24hrs
* How many patients on arrival were deemed to be unnecessary

The nurses and physicians who are communicating with the Intensivist about the case will complete a post-encounter survey to evaluate their experience.

ELIGIBILITY:
Remote Technology Group Inclusion:

* Patients ≤ 17 years from peripheral centre (Pelican Narrows Clinic and Regina General Hospital).
* Acutely ill.
* Being considered for medical transport.

Control Group Inclusion:

* Patients ≤ 17 years from peripheral centre (Stony Rapids, Wollaston Lake and Sandy Bay).
* Chosen from a pre-existing Saskatchewan paediatric transport database.

Exclusion Criteria:

* Patients older than age 17.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2015-03; Primary Completion 2016-02 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Transport number in the cases (with the robot) versus the controls (without the robot) | One year

SECONDARY OUTCOMES:
Tertiary care hospital length of stay in the cases versus the controls | One year
The number of patients transported to the regional hospitals in the cases (with the robot) versus the controls (without the robot) | One year

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Holt, MD, Principal Investigator — Clinical Assistant Professor
Locations (3):
- Canada (3):
  - Pelican Narrows Clinic (Angelique Canada Health Centre), Pelican Narrows, Saskatchewan
  - Regina General Hospital, Regina, Saskatchewan
  - Royal University Hospital, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Orr RA, Felmet KA, Han Y, McCloskey KA, Dragotta MA, Bills DM, Kuch BA, Watson RS. Pediatric specialized transport teams are associated with improved outcomes. Pediatrics. 2009 Jul;124(1):40-8. doi: 10.1542/peds.2008-0515. PMID 19564281
- [Background] Stroud MH, Prodhan P, Moss MM, Anand KJ. Redefining the golden hour in pediatric transport. Pediatr Crit Care Med. 2008 Jul;9(4):435-7. doi: 10.1097/PCC.0b013e318172da62. PMID 18496407
- [Background] Borrows EL, Lutman DH, Montgomery MA, Petros AJ, Ramnarayan P. Effect of patient- and team-related factors on stabilization time during pediatric intensive care transport. Pediatr Crit Care Med. 2010 Jul;11(4):451-6. doi: 10.1097/PCC.0b013e3181e30ce7. PMID 20453701
- [Background] Han YY, Carcillo JA, Dragotta MA, Bills DM, Watson RS, Westerman ME, Orr RA. Early reversal of pediatric-neonatal septic shock by community physicians is associated with improved outcome. Pediatrics. 2003 Oct;112(4):793-9. doi: 10.1542/peds.112.4.793. PMID 14523168
- [Background] Mendez I, Song M, Chiasson P, Bustamante L. Point-of-Care Programming for Neuromodulation: A Feasibility Study Using Remote Presence. Neurosurgery. 2013 Jan;72(1):99-108; discussion 108. doi: 10.1227/NEU.0b013e318276b5b2. PMID 23096417
- [Background] Rothenberg SS, Yoder S, Kay S, Ponsky T. Initial experience with surgical telementoring in pediatric laparoscopic surgery using remote presence technology. J Laparoendosc Adv Surg Tech A. 2009 Apr;19 Suppl 1:S219-22. doi: 10.1089/lap.2008.0133.supp. PMID 18976120